CLINICAL TRIAL: NCT00150735
Title: A Multicenter, Double-blind, Randomized, Parallel Group, Positive-controlled Trial Comparing the Efficacy and Safety of Levetiracetam (1000 to 3000 mg/Day Oral b.i.d.) to Carbamazepine (400 to 1200 mg/Day Oral b.i.d.), Used as Monotherapy for up to a Maximum of 121 Weeks in Subjects (≥ 16 Years) Newly or Recently Diagnosed as Suffering From Epilepsy, and Experiencing Partial or Generalized Tonic-clonic Seizures
Brief Title: Monotherapy With Levetiracetam in Newly Diagnosed Patients Suffering From Epilepsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: Double
Other Study IDs: N01061
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2010-07

CONDITIONS: Generalized Epilepsy
Keywords: Monotherapy, epilepsy, Levetiracetam, Keppra.
MeSH Terms: conditions — Epilepsy, Generalized; Epilepsy | interventions — Levetiracetam

INTERVENTIONS:
Drug: LEVETIRACETAM

SUMMARY:
A double-blind trial comparing the efficacy and safety of levetiracetam to carbamazepine used as monotherapy in subjects (≥ 16 years) newly or recently diagnosed as suffering from epilepsy, and experiencing partial or generalized tonic-clonic seizures.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with newly or recently diagnosed epilepsy having experienced unprovoked partial seizures (IA, IB, IC with clear focal origin), or generalized tonic-clonic seizures (without clear focal origin), that are classifiable according to the International Classification of Epileptic Seizures. The discrimination between IC and IIE is not requested for inclusion.
* Subjects with at least 2 unprovoked seizures separated by a minimum of 48 hours in the year preceding randomization out of which at least 1 unprovoked seizure in the 3 months preceding randomization.
* Subjects with a confirmed diagnosis of epilepsy.
* Male/female subjects (≥16 years).

Exclusion Criteria:

* History or presence of seizures of other types than partial (IA, IB, IC, with clear focal origin) and generalized tonic-clonic (without clear focal origin) seizures.
* History or presence of seizures occurring only in clustered patterns, defined as repeated seizures occurring over a short period of time, i.e. < 20 minutes, with or without function regained between 2 ictal events.
* History, clinical or EEG finding suggestive of idiopathic generalized epilepsy (IGE) at randomization.

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 580
Dates: Start 2002-06; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
To demonstrate that levetiracetam monotherapy is not inferior to carbamazepine by measuring the proportion of subjects with 6-month seizure freedom in subjects newly diagnosed as suffering from epilepsy.

SECONDARY OUTCOMES:
Proportion of subjects with one year seizure freedom; time to first seizure; safety.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma

REFERENCES:
- [Result] Brodie MJ, Perucca E, Ryvlin P, Ben-Menachem E, Meencke HJ; Levetiracetam Monotherapy Study Group. Comparison of levetiracetam and controlled-release carbamazepine in newly diagnosed epilepsy. Neurology. 2007 Feb 6;68(6):402-8. doi: 10.1212/01.wnl.0000252941.50833.4a. PMID 17283312